CLINICAL TRIAL: NCT01102543
Title: Observational Study in Neonatal Intensive Care Units (NICU) on the Real Life Use of Curosurf in Prophylaxis of RDS in Premature Babies.
Brief Title: Observational Study on the Prophylactic Use of Curosurf in Neonatal Respiratory Distress Syndrome (RDS)
Status: Completed | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CUR7101
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: pulmonary surfactant; Respiratory distress syndrome; Newborn; prophylaxis
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Premature babies < 28 GA
- Premature babies > 28 & < 32 weeks GA

SUMMARY:
The aim of Alizé is to describe a population of premature babies (gestational age (GA) < 32 weeks) in real life situation and the management of RDS.

DETAILED DESCRIPTION:
Description includes gestational age, birth clinical characteristics in particular the respiratory function, evaluation of the mother prenatal corticosteroids treatment in prophylaxis of RDS, mother medical and obstetric history, premature babies care in the delivery room with a special focus on the Curosurf use: prophylactic or curative use / other surfactant / no surfactant. A special focus is on the Prophylactic use.

ELIGIBILITY:
Inclusion Criteria:

* during the study, each neonatologist will have to include all the babies born with a gestational age < 32 GA

Exclusion Criteria:

* gestational age > 32 GA
* No consent to the data collection by one of the parents

Ages: 1 Minute to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 900 premature babies in 2 groups/cohorts : group 1 - babies born before 28 weeks GA ; groupe 2 - babies born at 28 - 32 weeks GA
Sampling Method: Probability Sample
Enrollment: 972 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Capucine de Meynard, MD, Study Director — Chiesi S.A.
Locations (1):
- Laboratoire Chiesi S.A., Courbevoie, France